CLINICAL TRIAL: NCT00280332
Title: A Follow-up Colonoscopy Examination in Patients Who Had Previously Undergone Screening Colonoscopy
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Dr WK Leung, Chinese University of Hong Kong
Other Study IDs: FUC
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Colonic Cancer
Keywords: colonic adenoma, colonic advanced neoplasm
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: colonic adenoma
  Interventions: Procedure: colonoscopy
- B: colonic without adenoma
  Interventions: Procedure: colonoscopy

INTERVENTIONS:
Procedure: colonoscopy — proform a follow up colonoscopy in the 5 year period from index colonoscopy
  Other Names: follow up colonoscopy

SUMMARY:
* To determine the prevalence of colonic neoplasm in patients who had previously undergone screening colonoscopy
* To determine the optimal time interval for re-screening in average risk individuals
* To determine potential baseline characteristics that predicts adenoma recurrence

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second commonest cancer in Hong Kong, and tends to be increasing. Screening for colorectal cancer can reduce the cancer incidence and mortality by detecting early lesions. However, the best interval for a follow up colonoscopy, particularly for those with normal baseline colonoscopy, remains largely unknown.

This study aim to determine the prevalence of colonic neoplasm in average-risk patients who had previously undergone screening colonoscopy and the optimal time interval for re-screening.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are previously participated in one of our two screening colonoscopy studies [Sung, Gastroenterol 2003; Leung, AJG 2004]
* Asymptomatic on first screening colonoscopy
* Age>50and <75
* No family history of CRC
* No other colonoscopy except the baseline screening colonoscopy

Exclusion Criteria:

* Subjects who refused consent
* Subjects who are not warrant follow up colonoscopy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who are previously participated in one of our two screening colonoscopy studies [Sung, Gastroenterol 2003; Leung, AJG 2004]
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2006-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The prevalence of advanced colonic adenoma in the re-screening population | 5 year from index colonoscopy

SECONDARY OUTCOMES:
The time to adenoma adenoma development according to different baseline characteristics of patients and colonoscopy findings | 5 years from index colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Wai K Leung, MD, Principal Investigator — CUHK
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong (sar), China